CLINICAL TRIAL: NCT05116163
Title: Breaking Implicit Bias Habits: An Individuation Pilot to Promote Equity in Rheumatic Disease Care
Brief Title: Breaking Implicit Bias Habits: An Individuation Pilot Study In Rheumatology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Virginia Commonwealth University (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Candace Hillary Feldman, MD, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021P002882; 5P30AG064199 (NIH)
Record Dates: First submitted 2021-10-13; First posted 2021-11-10 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Systemic Lupus Erythematosus; Rheumatoid Arthritis; Inflammatory Arthritis; Osteoarthritis
Keywords: Implicit Bias; Quality of Care; Rheumatology
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Arthritis; Osteoarthritis; Bias, Implicit

STUDY DESIGN:
Intervention Model Description: The investigators plan to enroll 20 rheumatologists and a maximum of 200 patients randomized into two different control arms. The providers will observe the outcomes in each separate arm as well as evaluate the results of both arms to each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Individuation Intervention plus implicit bias education (Experimental): 10 rheumatologists who will have 10 patient interactions each (100 patients total) recorded Rheumatologists will watch implicit bias training modules and then will be instructed to incorporate an individuation strategy into each of their clinical encounters.
  Interventions: Behavioral: Individuation Intervention plus implicit bias educational modules; Other: Implicit bias educational modules
- Arm 2: Implicit bias education only (Active Comparator): 10 rheumatologists randomized and stratified by hospital and gender
  Interventions: Other: Implicit bias educational modules

INTERVENTIONS:
Behavioral: Individuation Intervention plus implicit bias educational modules — Providers in the intervention are will be instructed to watch a brief set of freely available educational lessons and then they will meet with study team members to discuss their "individuation" countermeasure intervention. Providers will be given a choice of several individuation-related questions to better understand the unique characteristics of each patient. Once the provider decides on his/her choice phrases, the research team will assist with the development of a smart phrase (also called "dot phrase") to allow them to incorporate this into a note. Once a week, providers in the intervention arm will receive an email reminding them to incorporate this question and the documentation into their encounters.
  Arms: Arm 1: Individuation Intervention plus implicit bias education
Other: Implicit bias educational modules — Providers in the comparator arm will be given the same implicit bias educational modules to complete.

SUMMARY:
The first aim of this study is to test the efficacy of a real-time provider-based individuation intervention to improve the receipt of high-quality rheumatic disease care among Black/African American and lower socioeconomic status (SES) individuals. The second aim is to determine the effect of the individuation intervention on provider-patient communication, adherence, provider trust and care satisfaction.

DETAILED DESCRIPTION:
The goal of this pilot is to test the efficacy of an individuation-based intervention among rheumatologists and their patients at two large, multisite academic-based hospital practices to improve racial and SES equity in receipt of high quality care. The primary aim is not to reduce provider bias, but rather to reduce the reliance on implicit bias in care decisions for Black and lower SES patients to lessen the impact of structural racism and inequality on care.

The investigators plan to conduct a cluster-randomized controlled trial. The clusters are 20 rheumatologists at multisite BWH and MGH-affiliated clinics. Rheumatologists will be stratified by hospital and by gender and randomly assigned to one of two groups. Ten rheumatologists will be assigned to the intervention arm and ten to the control. Assessments will be conducted for 8-10 patients per rheumatologist (max 100 patients total in each arm, 200 total). Randomization will be stratified by BWH and MGH Rheumatology main campus hospitals (MGH or BWH/ Faulkner (FH)) and their rheumatology satellite clinic sites, and by provider gender (male or female). Inclusion and exclusion criteria for providers and patients are listed under Eligibility Criteria.

Providers who consent will be stratified by gender and site and randomized to the intervention or control arm. All providers in both arms will be asked to complete demographic surveys and four Implicit Association Tests (IATs). Two of the tests assess biases related to race and two parallel tests assess biases related to socioeconomic status. After providers take the IATs and complete the baseline demographics form, both arms will be given the link to freely available brief unconscious bias training module. The module that will be used has been approved by the MA Medical Society and is eligible for CME, which can be applied towards the unconscious bias training CMEs required for MA medical license renewal as of June 1, 2022. Upon completion of the unconscious bias module, providers in the intervention arm will meet with study team members to discuss their "individuation" countermeasure intervention and to view the brief presentation with a study team member about individuation.

At least one month after providers take the IATs, the study team will begin the process of recording 8-10 provider-patient interactions within each providers' practice. This will occur both at MGH and BWH rheumatology clinic sites. Providers will also be immediately informed before a patient encounter that will be recorded and will have the opportunity to decline. To record, a digital voice recorder will be used (placed in the room by a research team member with both patient and provider aware, and collected immediately following the encounter), and all data will be transferred to the project-specific MGB secure drive at the end of each day and then deleted from the device. These files will be transcribed verbatim using an MGB-approved vendor and all identifiable information will be removed. After 6 months, which is the estimate for recruitment time, providers will be asked to repeat the IATs.

Patients who consent to participate will be asked to have one clinical encounter with their provider recorded (preferably the next appointment) and then to complete a set of baseline surveys following that encounter including demographics, social determinants of health, everyday discrimination experiences, satisfaction with care, patient trust in the medical profession, patient perception of care centeredness and medication adherence. The investigators will also collect data from the patients' charts. These data include: demographics, social determinants of health, comorbidities/diagnoses, quality metrics related to their rheumatic disease, lab results, preventive care use (including immunizations), healthcare utilization (including ED visits, hospitalizations, outpatient visits and appointment no shows), medication use (including use of contraception as a quality metric), and medication refill data over the 6 months following the date of the recorded encounter. The investigators will review the note from the date of the encounter and determine whether the individuation statement was documented in the intervention group.

For patients with lupus, osteoarthritis, inflammatory arthritis, or RA seen at least once by participating providers in both the intervention and control arm, the study team will examine the charts of patients during the 6 months following provider enrollment, beginning 1 month after the date the provider takes the IATs. The study teams estimates that this will include approximately 1000 patients. The study team plan to collect demographics, social determinants of health, comorbidities/diagnoses, quality metrics related to their rheumatic disease, lab results, preventive care use (including immunizations), healthcare utilization (including ED visits, hospitalizations, outpatient visits and appointment no shows), medication use (including use of contraception as a quality metric), and medication refill data over the 6 months following the date of the recorded encounter. The investigators will also see if any of the individuation statements (smart phrases) were used for patients not specifically enrolled in the intervention.

At the end of the study, all data will be deidentified and analyzed in aggregate. Results in aggregate will be presented in an end-of-study Grand Rounds to both the BWH and MGH rheumatology divisions (there is a combined grand rounds). The team will also provide a list of online resources about implicit bias. For patients, after the completion of the 3-month adherence assessment, the study team will provide them with a score report indicating what their scores on each of the respective surveys mean.

ELIGIBILITY:
Inclusion Criteria:

* Providers: Providers will be male or female adult rheumatologists with >=1 clinical sessions/week at BWH/FH or MGH main campus and satellite clinic sites. The providers will aim to include a range of provider ages and years in practice.
* Patients: The study team will include male and female patients of the participating providers who are able to provide consent, English-speaking, >=18 years old, Black or African American or insured by Medicaid/Mass Health (as a proxy for low socioeconomic status), have a diagnosis of SLE, osteoarthritis, or inflammatory arthritis which includes RA (or referred to rheumatology because of high suspicion for these conditions), and have been seen <2 times in the past year by the provider.

Exclusion Criteria:

* Providers: Drs. Feldman and Schoenfeld (and their respective patients) will be excluded from this study.
* Patients: The providers will exclude patients who incarcerated or unable to consent. The providers will exclude any patient from our searches who has opted out of research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candace H Feldman, MD, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Rheumatologists were recruited from 6/17/2022-12/12/2023 at Brigham and Women's Hospital and Massachusetts General Hospital.
Pre-assignment Details: Rheumatologists took Implicit Association Tests and were provided with implicit bias training and then randomized to either the control or intervention arm.
Groups:
- Arm 1: Rheumatologist Individuation Intervention Plus Implicit Bias Education: Rheumatologists were randomized to this arm. They first watched implicit bias educational modules and then were instructed to incorporate an individuation strategy into each of their clinical encounters. Rheumatologists were given a choice of several individuation-related questions to better understand the unique characteristics of each patient. Once the provider decided on his/her choice phrases, the research team assisted with the development of a smart phrase (also called "dot phrase") to allow them to incorporate this into a note. Once a week, rheumatologists received an email reminding them to incorporate this question and the documentation into their encounters.
- Arm 2: Rheumatologist Implicit Bias Education Only: Rheumatologists were randomized to this arm. They watched implicit bias educational modules (same as those used in Arm 1) and received no further intervention.
- Patients of Arm 1 Providers- Chart Review Only: Patients of providers randomized to Arm 1 (individuation intervention). These patients were not intervened upon; their charts from routine care were reviewed only if they met inclusion criteria.
- Patients of Arm 2 Providers- Chart Review Only: Patients of providers randomized to Arm 2. These patients were not intervened upon; their charts from routine care were reviewed only if they met inclusion criteria.
- Patients of Arm 1 Rheumatologists Enrolled for Audiorecording: Patients of rheumatologists randomized to Arm 1 who consented for audiorecording and completed surveys, and participated in chart reviews.
- Patients of Arm 2 Rheumatologists Enrolled for Audiorecording: Patients of rheumatologists randomized to Arm 2 who consented for audiorecording and completed surveys, and participated in chart reviews.
Period: Overall Study
Arm/Group | Arm 1: Rheumatologist Individuation Intervention Plus Implicit Bias Education | Arm 2: Rheumatologist Implicit Bias Education Only | Patients of Arm 1 Providers- Chart Review Only | Patients of Arm 2 Providers- Chart Review Only | Patients of Arm 1 Rheumatologists Enrolled for Audiorecording | Patients of Arm 2 Rheumatologists Enrolled for Audiorecording
Started | 10 | 9 | 81 | 54 | 20 | 27
Completed | 10 | 9 | 79 | 50 | 19 | 27
Not Completed | 0 | 0 | 2 | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Rheumatologists and patients
Groups:
- Arm 1: Individuation Intervention Plus Implicit Bias Education: Rheumatologists: Rheumatologists watched implicit bias training modules and then were instructed to incorporate an individuation strategy into each of their clinical encounters.
- Arm 2: Implicit Bias Education Only: Rheumatologists: Rheumatologists watched implicit bias training modules.
- Patients of Arm 1- Chart Review Only: Patients of providers in Arm 1 who had their electronic health records reviewed but did not enroll/complete surveys
- Patients of Arm 2- Chart Review Only: Patients of providers in Arm 2 who had their electronic health records reviewed but did not enroll/complete surveys
- Patients of Arm 1 Providers With Audiorecordings and Surveys: Patients of providers in Arm 1 who enrolled for an audiorecorded encounter and surveys
- Patients of Arm 2 Providers With Audiorecordings and Surveys: Patients of providers in Arm 2 who enrolled for an audiorecorded encounter and surveys
- Total: Total of all reporting groups
Arm/Group | Arm 1: Individuation Intervention Plus Implicit Bias Education: Rheumatologists | Arm 2: Implicit Bias Education Only: Rheumatologists | Patients of Arm 1- Chart Review Only | Patients of Arm 2- Chart Review Only | Patients of Arm 1 Providers With Audiorecordings and Surveys | Patients of Arm 2 Providers With Audiorecordings and Surveys | Total
Number analyzed (Participants) | 10 | 9 | 79 | 50 | 20 | 27 | 195
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 53 | 38 | 17 | 23 | 148
  >=65 years | 1 | 1 | 26 | 12 | 3 | 4 | 47
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 5 | 5 | 53 | 37 | 11 | 17 | 128
  Male | 5 | 4 | 6 | 4 | 4 | 2 | 25
  Unknown | 0 | 0 | 20 | 9 | 5 | 8 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 9 | 10 | 2 | 5 | 29
  Not Hispanic or Latino | 9 | 6 | 67 | 38 | 17 | 21 | 158
  Unknown or Not Reported | 1 | 0 | 3 | 2 | 1 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 2 | 0 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 61 | 37 | 14 | 23 | 136
  White | 8 | 6 | 10 | 6 | 3 | 4 | 37
  More than one race | 0 | 0 | 2 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 1 | 0 | 6 | 5 | 2 | 0 | 14
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 79 | 50 | 20 | 27 | 248
Provider-Only Implicit Association Test- Race Bias [Mean (Standard Deviation); unit: units on a scale] — Implicit Association Test for Black/White racial implicit bias completed by rheumatologists only. The score ranges from -2 to +2 where -2 indicates pro-Black bias and +2 indicates pro-White bias. A score of 0 indicates no preference. Population: This analysis was only completed for providers; therefore the number analyzed for each of the patient categories is 0.
  units on a scale
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 0 | 0 | 19
    (all) | -0.46 (0.54) | -0.37 (0.57) |  |  |  |  | -0.42 (0.54)
Provider-Only Implicit Association Tests - Race stereotyping [Mean (Standard Deviation); unit: units on a scale] — Implicit Association Tests for Black/White race stereotyping completed by providers only. The score ranges from -2 to +2 where -2 indicates pro-Black stereotyping and +2 indicates pro-White stereotyping. A score of 0 indicates no preference. Population: Provider only surveys
  units on a scale
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 0 | 0 | 19
    (all) | -0.13 (0.76) | -0.29 (0.37) |  |  |  |  | -0.20 (0.60)
Provider-Only Implicit Association Test - Socioeconomic status bias [Mean (Standard Deviation); unit: units on a scale] — Implicit association tests for high vs. low socioeconomic status bias completed by providers only. The score ranges from -2 to +2 where -2 indicates pro-low SES bias and +2 indicates pro-high SES bias. A score of 0 indicates no preference. Population: Provider only surveys
  units on a scale
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 0 | 0 | 19
    (all) | 0.75 (0.55) | 0.54 (0.35) |  |  |  |  | 0.65 (0.47)
Provider-Only Implicit Association Test - Socioeconomic status stereotyping [Mean (Standard Deviation); unit: units on a scale] — Implicit association test for high vs. low socioeconomic status stereotyping completed by providers only. The score ranges from -2 to +2 where -2 indicates pro-low SES stereotyping and +2 indicates pro-high SES stereotyping. A score of 0 indicates no preference. Population: Provider only surveys
  units on a scale
    number analyzed (Participants) | 10 | 9 | 0 | 0 | 0 | 0 | 19
    (all) | 0.54 (0.60) | 0.48 (0.49) |  |  |  |  | 0.51 (0.54)
Baseline Medication Adherence [Mean (Standard Deviation); unit: units on a scale] — Baseline three-question measure of medication adherence with a mean calculated across the three items and a range of 0-100. Higher scores indicate greater adherence. Population: Enrolled patient-only measure
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 20 | 27 | 47
    (all) |  |  |  |  | 49.3 (19.6) | 58.9 (18.8) | 53.8 (19.5)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Quality Metrics Achieved
Description: Documented receipt of high-quality care at the appointment or within 30 days of the appointment. The quality metrics for Lupus and RA include but are not limited to: Hydroxychloroquine (HCQ) initiation and Folic acid if receiving methotrexate, respectively. These items will be added together to form a score and the number of items completed out of the total will be the primary outcome measure compared across groups. The denominator is the patient-specific quality metrics they are eligible for and the numerator is the number achieved. The final percent ranges from 0-100 (with 100 indicating that 100% of the quality metrics that the patient was eligible for were met).
Time Frame: 30 days
Population: Patients of providers randomized to Arm 1 or Arm 2, which includes the eligible patients in the chart-review groups, and those who also participated in the audiorecordings and surveys
Measure: Mean (Standard Deviation); unit: Percent of Quality Metrics Achieved
Groups:
- Patients of Arm 1 Providers; Patients of Arm 2 Providers: Includes all patients in the chart review arm and in the audiorecording/survey arms.
Arm/Group | Patients of Arm 1 Providers | Patients of Arm 2 Providers
Number analyzed (Participants) | 98 | 77
Percent of Quality Metrics Achieved | 62.14 (13.46) | 54.31 (14.46)
Statistical Analysis 1: Comparison: Patients of Arm 1 Providers vs Patients of Arm 2 Providers; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 7.83, Standard Error of Mean 2.05 — Difference in the mean of percent of quality metrics achieved in the intervention arm minus the control arm

2. Secondary Outcome: Perception of Patient Centeredness
Description: Differences in perception of patient centeredness comparing the intervention to non-intervention group. Higher scores indicate less patient-centered experiences. 4-point Likert scale, score range from 14-56.
Time Frame: At time of appointment (baseline) during which audiorecording took place, reflecting the experience at the appointment immediately preceding survey completion.
Population: Subset of patients who consented to participate in audiorecordings and returned completed surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys: Subset of patients of providers in Arm 1 who enrolled for audiorecordings and completed surveys
- Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys: Subset of patients of providers in Arm 2 who enrolled in audiorecording and completed surveys
Arm/Group | Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys | Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys
Number analyzed (Participants) | 19 | 21
score on a scale | 27.5 (9) | 23.4 (7)
Statistical Analysis 1: Comparison: Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys vs Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys; Test type: Superiority; p = 0.1164, t-test, 2 sided; Mean Difference (Final Values) = 4.1

3. Secondary Outcome: Patient Satisfaction
Description: Differences in patient satisfaction score, comparing the intervention to non-intervention group. Score range from 20-70. Higher scores indicate greater patient satisfaction.
Time Frame: as for outcome 2
Population: Subset of patients who consented to participate in audiorecordings and returned completed surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys | Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys
Number analyzed (Participants) | 17 | 22
score on a scale | 50.4 (9) | 51.5 (8)
Statistical Analysis 1: Comparison: Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys vs Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys; Test type: Superiority; p = 0.6781, t-test, 2 sided; Mean Difference (Final Values) = -1.1 — Intervention group mean - control group mean

4. Secondary Outcome: Everyday Discrimination Scale
Description: Reflects experiences of everyday discrimination, comparing the intervention to non-intervention group. Score range is 0-40. Higher scores indicate a greater amount of discrimination encountered.
Time Frame: A time of the appointment when audiorecording took place (baseline) asking patients to describe the degree to which each item occurs in their day-to-day life.
Population: Subset of patients who consented to participate in audiorecordings and returned completed surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys | Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys
Number analyzed (Participants) | 19 | 25
score on a scale | 0.96 (0.84) | 1.16 (0.93)
Statistical Analysis 1: Comparison: Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys vs Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys; Test type: Superiority; p = 0.4795, t-test, 2 sided; Mean Difference (Final Values) = -0.2 — Intervention group mean - control group mean

5. Secondary Outcome: Adherence
Description: Adherence score (for rheumatology medications), comparing the 3-month adherence score to baseline for the intervention to non-intervention group at three months following the encounter date. Score range is 0-100 with zero being the lowest adherence, and 100 being the best.
Time Frame: 3 months after the start of the intervention
Population: Subset of patients in the audiorecording/survey arms who returned completed 3 month follow up adherence surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys | Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys
Number analyzed (Participants) | 13 | 12
score on a scale | 54.96 (14.15) | 55.99 (19.44)
Statistical Analysis 1: Comparison: Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys vs Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys; Comparison of 3-month vs. baseline adherence scores in patients of providers in the intervention arm vs. control; Test type: Superiority; p = 0.056, Regression, Linear

6. Secondary Outcome: Provider Communication: Positive Emotion Words
Description: Provider communication will be measured using the recorded transcripts and compared between arms. We compared the mean (SD) of provider positive emotion words expressed during a clinical encounter. Measured only for patients enrolled in the study who had their appointment audiorecorded.
Time Frame: One time baseline evaluation from the transcript of the audiorecording of the encounter of the patient with their rheumatologist
Population: Patients who participated in audiorecordings and had transcripts for analysis.
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys | Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys
Number analyzed (Participants) | 19 | 27
Number of words | 0.99 (0.50) | 0.66 (0.33)
Statistical Analysis 1: Comparison: Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys vs Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys; Test type: Superiority; p = 0.017, t-test, 2 sided; Mean Difference (Final Values) = 0.33

7. Secondary Outcome: Patient Trust
Description: Patient trust in their providers, comparing the intervention to non-intervention group. Responses are summed (range 5-25) with higher scores indicating more trust.
Time Frame: One time baseline evaluation after the appointment reflecting experiences at the immediately preceding appointment.
Population: Subset of patients who consented to participate in audiorecordings and returned completed surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys | Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys
Number analyzed (Participants) | 19 | 24
score on a scale | 16.4 (4) | 17.6 (5)
Statistical Analysis 1: Comparison: Patients of Arm 1 Providers Enrolled for Audiorecording and Surveys vs Patients of Arm 2 Providers Enrolled for Audiorecording and Surveys; Test type: Superiority; p = 0.3957, t-test, 2 sided; Mean Difference (Final Values) = -1.2 — Mean from intervention arm - control arm

8. Secondary Outcome: Incidence Rate Ratio of Emergency Departments Visits
Description: Comparison of incidence rate of Emergency Department visits between patients of providers in the intervention compared to the control arms.
Time Frame: 6 months following the encounter of interest
Measure: Mean (Standard Deviation); unit: number of ED visits
Groups:
- Patients of Arm 1 Providers; Patients of Arm 2 Providers: Includes all patients in the chart review arm (which also includes the subarm that had audiorecorded encounters and completed surveys)
Arm/Group | Patients of Arm 1 Providers | Patients of Arm 2 Providers
Number analyzed (Participants) | 98 | 77
number of ED visits | 0.398 (0.971) | 0.390 (0.934)
Statistical Analysis 1: Comparison: Patients of Arm 1 Providers vs Patients of Arm 2 Providers; Comparing the incidence rate of ED visits for the intervention vs. control arms; Test type: Superiority; Incidence Rate Ratio = 1.02, 95% CI 2-sided [0.63 to 1.64]

9. Secondary Outcome: Incidence Rate Ratio of Outpatient Visits.
Description: Comparison of incidence rate of outpatient visits between patients of providers in the intervention compared to the control arms.
Time Frame: 6 months following the encounter of interest
Measure: Mean (Standard Deviation); unit: Number of outpatient visits
Arm/Group | Patients of Arm 1 Providers | Patients of Arm 2 Providers
Number analyzed (Participants) | 98 | 77
Number of outpatient visits | 7.34 (6.22) | 6.05 (5.88)
Statistical Analysis 1: Comparison: Patients of Arm 1 Providers vs Patients of Arm 2 Providers; Incidence rate ratio comparing incidence rates of outpatient visits in the intervention vs. control arms; Test type: Superiority; Incidence Rate Ratio = 1.21, 95% CI 2-sided [1.07 to 1.36]

10. Secondary Outcome: Incidence Rate Ratio of Hospitalizations
Description: Comparison of incidence rate of hospitalizations between patients of providers in the intervention compared to the control arms.
Time Frame: 6 months after physician encounter
Measure: Mean (Standard Deviation); unit: number of hospitalizations
Arm/Group | Patients of Arm 1 Providers | Patients of Arm 2 Providers
Number analyzed (Participants) | 98 | 77
number of hospitalizations | 0.316 (1.06) | 0.779 (0.354)
Statistical Analysis 1: Comparison: Patients of Arm 1 Providers vs Patients of Arm 2 Providers; Incidence rate ratio comparing the incidence rates of hospitalizations in the intervention vs. control arm patients; Test type: Superiority; Incidence Rate Ratio = 4.06, 95% CI 2-sided [1.69 to 9.73]

11. Secondary Outcome: Implicit Association Test (IAT) Scores- Socioeconomic Status Stereotyping
Description: Change in provider IAT scores pre and post intervention. IAT scores range from -1 to 1. A score of 0 indicates no strong implicit bias. A score of 1 is pro-high socioeconomic status bias and a score of -1 is pro-low socioeconomic status bias.
Time Frame: Baseline compared to 6 months after the start of the intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Individuation Intervention Plus Implicit Bias Education: Rheumatologists who will have 10 patient interactions each (100 patients total) recorded Rheumatologists will watch implicit bias training modules and then will be instructed to incorporate an individuation strategy into each of their clinical encounters.
  Individuation Intervention plus implicit bias educational modules: Providers in the intervention are will be instructed to watch a brief set of freely available educational lessons and then they will meet with study team members to discuss their "individuation" countermeasure intervention. Providers will be given a choice of several individuation-related questions to better understand the unique characteristics of each patient. Once the provider decides on his/her choice phrases, the research team will assist with the development of a smart phrase (also called "dot phrase") to allow them to incorporate this into a note. Once a week, providers in the intervention arm will receive an email reminding them to incorporate this question and the documentation into their encounters.
  Implicit bias educational modules: Providers in the comparator arm will be given the same implicit bias educational modules to complete.
- Arm 2: Implicit Bias Education Only: Rheumatologists randomized and stratified by hospital and gender
  Implicit bias educational modules: Providers in the comparator arm will be given the same implicit bias educational modules to complete.
Arm/Group | Arm 1: Individuation Intervention Plus Implicit Bias Education | Arm 2: Implicit Bias Education Only
Number analyzed (Participants) | 10 | 9
units on a scale | 0.50 (0.37) | 0.15 (0.50)
Statistical Analysis 1: Comparison: Arm 1: Individuation Intervention Plus Implicit Bias Education vs Arm 2: Implicit Bias Education Only; Post vs. pre IAT d-scores comparing the intervention vs. control arms; Test type: Superiority; p = 0.3882, t-test, 2 sided

12. Secondary Outcome: Implicit Association Test (IAT) Scores- Race Implicit Bias
Description: Change in provider IAT scores pre and post intervention. IAT scores range from -1 to 1. A score of 0 indicates no strong implicit bias. A score of 1 is pro-White bias and a score of -1 is pro-Black bias.
Time Frame: Baseline compared to 6 months after the start of the intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Individuation Intervention Plus Implicit Bias Education | Arm 2: Implicit Bias Education Only
Number analyzed (Participants) | 10 | 9
units on a scale | -0.27 (0.47) | 0.12 (0.44)
Statistical Analysis 1: Comparison: Arm 1: Individuation Intervention Plus Implicit Bias Education vs Arm 2: Implicit Bias Education Only; Comparing post vs. pre IAT d-scores between the intervention and control groups; Test type: Superiority; p = 0.3615, t-test, 2 sided

13. Secondary Outcome: Implicit Association Test (IAT) Scores- Race Stereotyping.
Description: Change in provider IAT scores pre and post intervention. IAT scores range from -1 to 1. A score of 0 indicates no strong implicit bias. A score of 1 is pro-White stereotyping and a score of -1 is pro-Black stereotyping.
Time Frame: Baseline compared to 6 months after the start of the intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Individuation Intervention Plus Implicit Bias Education | Arm 2: Implicit Bias Education Only
Number analyzed (Participants) | 10 | 9
units on a scale | -0.25 (0.61) | -0.39 (0.50)
Statistical Analysis 1: Comparison: Arm 1: Individuation Intervention Plus Implicit Bias Education vs Arm 2: Implicit Bias Education Only; Comparing post vs pre IAT d-scores in the intervention vs. control arms; Test type: Superiority; p = 0.9432, t-test, 2 sided

14. Secondary Outcome: Implicit Association Test (IAT) Scores- Socioeconomic Status Bias
Description: . Change in provider IAT scores pre and post intervention. IAT scores range from -1 to 1. A score of 0 indicates no strong implicit bias. A score of 1 is pro-high socioeconomic status bias and a score of -1 is pro-low socioeconomic status bias.
Time Frame: Baseline compared to 6 months after the start of the intervention.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1: Individuation Intervention Plus Implicit Bias Education | Arm 2: Implicit Bias Education Only
Number analyzed (Participants) | 10 | 9
units on a scale | 0.48 (0.37) | 0.60 (0.56)
Statistical Analysis 1: Comparison: Arm 1: Individuation Intervention Plus Implicit Bias Education vs Arm 2: Implicit Bias Education Only; Post vs pre IAT d-scores for the intervention vs. control arms; Test type: Superiority; p = 0.1453, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The study period was six months.
Description: The clinicaltrials.gov definitions were used.
Groups:
- Arm 1: Individuation Intervention Plus Implicit Bias Education: 10 rheumatologists will watch implicit bias training modules and then will be instructed to incorporate an individuation strategy into each of their clinical encounters.
  Individuation Intervention plus implicit bias educational modules: Providers in the intervention are will be instructed to watch a brief set of freely available educational lessons and then they will meet with study team members to discuss their "individuation" countermeasure intervention. Providers will be given a choice of several individuation-related questions to better understand the unique characteristics of each patient. Once the provider decides on his/her choice phrases, the research team will assist with the development of a smart phrase (also called "dot phrase") to allow them to incorporate this into a note. Once a week, providers in the intervention arm will receive an email reminding them to incorporate this question and the documentation into their encounters.
  Implicit bias educational modules: Providers in the comparator arm will be given the same implicit bias educational modules to complete.
- Patients of Arm 1 Providers- Chart Review Only: Patients of providers randomized to Arm 1 (individuation intervention). These patients were not enrolled; their charts were reviewed only.
- Patients of Arm 2 Providers- Chart Review Only: Patients of providers randomized to Arm 2 (education-only arm). These patients were not enrolled; their charts were reviewed only.
- Arm 1 Patients Enrolled for Audiorecording: Subset of chart reviewed patients of Arm 1 providers who consented for audiorecording and completed surveys.
- Arm 2 Patients Enrolled for Audiorecording: Subset of chart reviewed patients of Arm 2 providers who consented for audiorecording and completed surveys.
Arm/Group | Arm 1: Individuation Intervention Plus Implicit Bias Education | Arm 2: Implicit Bias Education Only | Patients of Arm 1 Providers- Chart Review Only | Patients of Arm 2 Providers- Chart Review Only | Arm 1 Patients Enrolled for Audiorecording | Arm 2 Patients Enrolled for Audiorecording
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/101 | 0/81 | 0/20 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/101 | 0/81 | 0/20 | 0/27
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/101 | 0/81 | 0/20 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT05116163/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT05116163/ICF_000.pdf